CLINICAL TRIAL: NCT02536248
Title: EFFECTS OF SITAGLIPTIN THERAPY ON THE KINETICS OF MARKERS OF LOW-GRADE INFLAMMATION AND CELL ADHESION MOLECULES IN PATIENTS WITH TYPE 2 DIABETES
Brief Title: Sitagliptin Therapy and Kinetics of Inflammatory Markers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Couture, MD, PhD, FRCP, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JANU-INF
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: sitagliptin; diabetes; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Inflammation | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin first, then Placebo (Experimental): Sitagliptin 100 mg/d for 6 weeks
  Wash-out 14 days
  Placebo for 6 weeks
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Placebo first, then Sitagliptin (Placebo Comparator): Placebo for 6 weeks
  Wash-out 14 days
  Sitagliptin 100 mg/d for 6 weeks
  Interventions: Drug: Sitagliptin; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg/d for 6 weeks
  Other Names: Januvia
Drug: Placebo — Placebo for 6 weeks

SUMMARY:
Inflammatory processes are increasingly being recognized as a critical step in the pathogenesis of both diabetes and heart disease and may constitute a biological link between the two diseases. Inflammatory cytokines increase vascular permeability, change vasoregulatory responses, increase leukocyte adhesion to endothelium, and facilitate thrombus formation by inducing procoagulant activity, inhibiting anticoagulant pathways, and impairing fibrinolysis. Leukocyte adhesion to arterial endothelial cells is thought to be an important step in the development of atherosclerosis, and adhesion molecules, such as intercellular adhesion molecule-1 (ICAM-1) and L-selectin, play key roles in this process. Therefore, identifying novel therapeutic approaches that would favorably affect inflammation, endothelial function, and glucose is of significant interest. Investigators have recently demonstrated that, relative to placebo, sitagliptin treatment resulted in a significant reduction in plasma levels of various inflammatory markers and cell adhesion molecules. The results also suggest that the beneficial effects of sitagliptin on both inflammation and endothelial function are most likely mediated by an elevation in plasma GLP-1 levels and global improvement of the glucose-insulin homeostasis. However, the mechanisms underlying the beneficial effects of sitagliptin on these markers remain to be fully elucidated. The proposed study will address this key issue.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 65 years of age.
* Post-menopausal women under age 65 on stable medical therapy for 6 months before the study (the patient should have demonstrated stable lipid panels)
* Women should not be on hormone replacement therapy (no recent starting or stopping)
* Type 2 diabetes as defined by the American Diabetes Association.
* Non-smoker.
* Body mass index between 25.0 and 40.0 kg/m2.
* Baseline glycated hemoglobin A1c (HbA1c) between 6.5 and 8.5%.
* Baseline fasting plasma glucose < 15.0 mmol/L.
* Plasma triglyceride levels between 1.5 and 8.0 mmol/L (135 and 710 mg/dl) at screening and week -4.
* Patients having received stable doses of metformin for at least 3 months before randomization.
* Subjects must be willing to give written informed consent and able to adhere to dosing schedule, visit schedule and phone follow-up assessment.
* Patients should be otherwise generally healthy, without elevations in hepatic transaminases or abnormal renal function or coagulation.
* Patients having normal thyroid stimulating hormone at screening

Exclusion Criteria:

* Patients with extreme dyslipidemias, such as familial hypercholesterolemia will be excluded.
* Patients with type 1 diabetes, secondary form of diabetes or acute metabolic diabetic complications will be excluded.
* Patients having received or being treated with insulin or a thiazolidinedione within the past 6 months will be excluded.
* Patients taking any other hypoglycemic agent, other than metformin.
* Subjects will be excluded if they have cardiovascular disease (coronary heart disease, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (e.g. steroids, beta blockers, thiazide diuretics, lipid lowering agents, significant alcohol intake etc.).
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Individuals with a history of mental instability, drug or alcohol abuse or individuals who have been treated or are being treated for severe psychiatric illness that, in the opinion of the investigator, may interfere with optimal participation in the study.
* History of alcohol or drug abuse within the past 2 years. Patients must not take alcohol during the study.
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease, that would limit study evaluation or participation.
* Known impairment of renal function (serum creatinine levels > 1.7 mg/dL for men), dysproteinemia, nephrotic syndrome, or other renal disease (24-hour urinary protein ≥3 ± 1 g).
* Active or chronic hepatobiliary or hepatic disease. In addition, patients with aspartate aminotransferase or alanine aminotransferase >2 x upper limit of the laboratory reference range will be excluded.
* Subjects with coagulopathy (prothrombin time or partial thromboplastin time at Visit 1 >1.5 times control).
* Subjects with hemoglobin >2 x the lower limit of the laboratory reference range will be excluded.
* Patients who are known to have tested positive for human immunodeficiency virus (HIV).
* Patients who are currently enrolled in another clinical study.
* Patients who have used any investigational drug within 30 days of the first clinic visit.
* Congestive heart failure New York Heart Association (NYHA) Class III or IV. Uncontrolled cardiac arrhythmias within 3 months of study entry.
* Uncontrolled diabetes mellitus (HbA1c>8.5%) or other endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid subjects on replacement doses of thyroid hormone are eligible for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, FRCP, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin First Then Placebo: Sitagliptin 100 mg/d for 6 weeks
  Wash-out 14 days
  Placebo for 6 weeks
Period: First Intervention (6 Weeks)
Arm/Group | Sitagliptin First Then Placebo | Placebo First, Then Sitagliptin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Wash-out (14 Days)
Arm/Group | Sitagliptin First Then Placebo | Placebo First, Then Sitagliptin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Sitagliptin First Then Placebo | Placebo First, Then Sitagliptin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin First Then Placebo: Sitagliptin 100 mg/d for 6 weeks
  Sitagliptin: Sitagliptin 100 mg/d for 6 weeks
- Placebo First Then Sitagliptin: Placebo for 6 weeks
  Placebo: Placebo for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Sitagliptin First Then Placebo | Placebo First Then Sitagliptin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (4.6) | 58.5 (3.2) | 58.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Measurement of C-reactive Protein Production Rate With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Population: Results for this outcome are not available since we had issues with the measurement of deuterated leucine in the current protein (C-reactive protein).
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Measurement of Serum Amyloid A Production Rate With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 20 | 20
mg/kg/day | 0.039 (0.030) | 0.049 (0.047)

3. Secondary Outcome: Measurement of L-selectin Production Rate With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Population: Results for this outcome are not available since we had issues with the measurement of deuterated leucine in the current protein (L-selectin).
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measurement of ICAM-1 Production Rate With Stable Isotope During Postprandial Period
Time Frame: 6 weeks
Population: Results for this outcome are not available since we had issues with the measurement of deuterated leucine in the current protein (I-CAM-1).
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During 16 weeks
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02536248/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02536248/SAP_001.pdf